CLINICAL TRIAL: NCT05142722
Title: A Placebo-Controlled, Double-Blind, Randomized Phase 3 Study to Evaluate the Effect of 10mg Obicetrapib in Participants With HeFH and/or ASCVD Who Are Not Adequately Controlled by Their Lipid Modifying Therapies
Brief Title: Randomized Study to Evaluate the Effect of Obicetrapib on Top of Maximum Tolerated Lipid-Modifying Therapies
Acronym: BROADWAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-302
Record Dates: First submitted 2021-11-18; First posted 2021-12-03 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-02

CONDITIONS: Dyslipidemias; High Cholesterol; Hypercholesterolemia; Familial Hypercholesterolemia; Atherosclerotic Cardiovascular Disease
Keywords: obicetrapib; BROADWAY; Cholesteryl ester transfer protein (CETP) inhibitor; Heterozygous Familial Hypercholesterolemia (HeFH); Atherosclerotic Cardiovascular Disease (ASCVD)
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hyperlipoproteinemia Type II; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo tablet made to resemble active
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): one placebo tablet once daily
  Interventions: Drug: Placebo
- obicetrapib 10mg (Experimental): one 10mg obicetrapib tablet once daily
  Interventions: Drug: Obicetrapib

INTERVENTIONS:
Drug: Placebo — placebo tablet made to resemble active
  Arms: Placebo
Drug: Obicetrapib — 10mg obicetrapib tablet
  Arms: obicetrapib 10mg

SUMMARY:
This study will be a placebo-controlled, double-blind, randomized, phase 3 study in participants with underlying heterozygous familial hypercholesterolemia (HeFH) and/or ASCVD to evaluate the efficacy, safety, and tolerability of obicetrapib as an adjunct to diet and maximally tolerated lipid-lowering therapy

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, randomized, phase 3 study in participants with underlying HeFH and/or ASCVD to evaluate the efficacy, safety, and tolerability of obicetrapib as an adjunct to diet and maximally tolerated lipid-lowering therapy. The screening period for this study will take up to 28 days. Afterwards patients will be randomized to placebo or 10 mg obicetrapib for a 365 day treatment period. After the treatment period, patients will have an end of study follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Females may be enrolled if all 3 of the following criteria are met:
* They are not pregnant;
* They are not breastfeeding; and
* They do not plan on becoming pregnant during the study;
* Have underlying heterozygous familial hypercholesterolemia (HeFH) and/or a history of established ASCVD
* Are on maximally tolerated lipid-modifying therapy as an adjunct to a lipid-lowering diet and other lifestyle modifications, defined as follows:
* A statin at a maximally tolerated stable dose for at least 8 weeks prior to Screening
* Atorvastatin 40 and 80 mg; and
* Rosuvastatin 20 and 40 mg;
* Ezetimibe with or without maximally tolerated statin for at least 8 weeks prior to Screening
* Bempedoic acid with a maximally tolerated statin for at least 8 weeks prior to Screening
* A PCSK-9 targeted therapy alone or in combination with other lipid-modifying therapy for at least 4 stable doses prior to Screening
* Have a fasting serum LDL-C at Screening as follows:
* Fasting serum LDL-C ≥ 55 to < 100 mg/dL (≥1.4 to <2.6 mmol/L) OR non-HDL-C ≥85 mg/dL (≥2.2 mmol/L) to < 130 mg/dL (<3.4 mmol/L) with at least 1 of the following risk enhancers at Screening;
* Recent MI (> 3 and < 12 months prior to Randomization);
* Type 2 diabetes mellitus;
* Current daily cigarette smoking;
* Age of > 60 years;
* High sensitivity C-reactive protein (hsCRP) ≥2.0 mg/L (≥19.0 nmol/L) at Screening or within 6 months prior to Screening
* Fasting triglycerides (TG) > 150 mg/dL (>1.7 mmol/L);
* Fasting lipoprotein (a) > 30 mg/dL (>70 nmol/L); and/or
* Fasting HDL-C < 40 mg/dL (<1.0 mmol/L); OR
* Fasting serum LDL-C ≥ 100 mg/dL (≥2.6 mmol/L) or non-HDL-C ≥130 mg/dL (≥3.4 mmol/L)
* Fasting triglyceride (TG) < 500 mg/dL (<5.7 mmol/L) at Screening; and
* Have an estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73m2 at Screening

Exclusion Criteria:

* New York Heart Association class III or IV heart failure or left ventricular ejection fraction < 30%;
* Hospitalized for heart failure within 5 years prior to Screening
* Major adverse cardiac event (MACE) within 3 months prior to Screening;
* Uncontrolled severe hypertension, defined as either systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg prior to Randomization;
* Formal diagnosis of homozygous familial hypercholesterolemia (HoFH);
* Active liver disease;
* HbA1c ≥10% or a fasting glucose ≥270 mg/dL (≥15.0 mmol/L) at Screening;
* Thyroid-stimulating hormone >1.5 X upper limit of normal (ULN) at Screening;
* Creatine kinase > 3 X upper limit of normal (ULN) at Screening;
* History of malignancy that required surgery (excluding local and wide local excision), radiation therapy, and/or systemic therapy during the 3 years prior to Randomization;
* Known history of alcohol and/or drug abuse within 5 years prior to Randomization
* Received treatment with other investigational products or devices within 30 days of Screening or 5 half-lives of the previous investigational product, whichever is longer;
* Are taking gemfibrozil or have taken gemfibrozil within 30 days of Screening
* Planned use of other investigational products or devices during the course of the study;
* Participated in any clinical trial evaluating obicetrapib; or
* Known allergy or hypersensitivity to obicetrapib, placebo, or any of the excipients in obicetrapib or placebo
* Any condition that, according to the Investigator, could interfere with the conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2530 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ditmarsch, Study Director — NewAmsterdam Pharma
Locations (181):
- United States (69):
  - Pinnacle Research Group, Anniston, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Synexus Clinical Research US, Inc. / Simon Williamson Clinic, PC, Birmingham, Alabama
  - The Center for Clinical Trials, Inc, Saraland, Alabama
  - Syed Research Consultants, LLC, Sheffield, Alabama
  - Clinical Research Institute of Arizona, LLC, Sun City West, Arizona
  - Synexus Clinical Research US, Inc. / Orange Grove Family Practice, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - American Institute of Research, Beverly Hills, California
  - Orange County Research Center, Tustin, California
  - Synexus Clinical Research US, Inc., Vista, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Pioneer Clinical Studies, Ft. Pierce, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - East Coast Institute for Research, LLC - Jacksonville University Blvd, Jacksonville, Florida
  - East Coast Institute for Research- Lake City, Lake City, Florida
  - ClinCloud LLC, Maitland, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Progressive Medical Research, Port Orange, Florida
  - East Coast Institute for Research, Saint Augustine, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - East Coast Institute for Research - Canton, Canton, Georgia
  - Centricity Research, Columbus, Georgia
  - East Coast Institute for Research, LLC, Macon, Georgia
  - Alta Pharmaceutical Research Center, Peachtree Corners, Georgia
  - SouthCoast Health, Savannah, Georgia
  - Biofortis, Inc, Addison, Illinois
  - Evanston Premier Healthcare Research LLC, Skokie, Illinois
  - Synexus Clinical Research US, Inc., Evansville, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Grace Research, LLC, Bossier City, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Tandem Clinical Research GI - Metairie, Metairie, Louisiana
  - Grace Research, LLC, Shreveport, Louisiana
  - Southern Clinical Research, LLC, Zachary, Louisiana
  - Northern Light Cardiology, Bangor, Maine
  - Privia Medical Group, LLC, Silver Spring, Maryland
  - Oakland Medical Research, Troy, Michigan
  - Arcturus Healthcare, Troy Internal Medicine Research Division, Troy, Michigan
  - AB Clinical Trials, Las Vegas, Nevada
  - Inspira Medical Centers dba Internal Medicine Associates, P.A., Bridgeton, New Jersey
  - Mid Hudson Medical Research, New Windsor, New York
  - Synexus Clinical Research US, Inc., New York, New York
  - Tandem Clinical Research GI, LLC, New York, New York
  - Chear Center LLC, The Bronx, New York
  - Diabetes and Endocrinology Consultants, P.C., Morehead City, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Summit Research Group, LLC, Stow, Ohio
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Cardiovascular Research of Knoxville, LLC, Powell, Tennessee
  - Amarillo Heart Clinical Research Institute, Inc, Amarillo, Texas
  - Inquest Clinical Research, Baytown, Texas
  - Apex Mobile Clinical Research, Bellaire, Texas
  - Javara Inc., Conroe, Texas
  - Prime Revival Research Institute, LLC, Coppell, Texas
  - Thyroid, Endocrinology & Diabetes, PA, Dallas, Texas
  - Northwest Houston Clinical Research, Tomball, Texas
  - Synexus Clinical Research US, Inc., Salt Lake City, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - Hampton Roads Center for Clinical Research, Suffolk, Virginia
  - Universal Research Group, LLC, Tacoma, Washington
- China (29):
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Cangzhou Central Hospital, Cangzhou
  - China-Japan Union Hospital Of Jilin University, Changchun
  - The First People's Hospital of Changde City, Changde
  - The Second People's Hospital of Changzhou, Changzhou
  - Affiliated Hospital of Chifeng University, Chifeng
  - Chifeng Municipal Hospital, Chifeng
  - Daqing People's Hospital, Daqing
  - Foshan First People's Hospital, Foshan
  - Guangdong Provincial People's Hospital, Guangzhou
  - The Third Affiliated Hospital of Guangzhou Medical university, Guangzhou
  - Heilongjiang Provincial Hospital, Harbin
  - The First Affiliated Hospital Of University Of South China, Hunan
  - Jinan Central Hospital, Jinan
  - Hebei Petro China Central Hospital, Langfang
  - Lishui Central Hospital, Lishui
  - Luoyang Third People's Hospital, Luoyang
  - The First affiliated Hospital of Nanyang Medical College, Nanyang
  - Panjin Liaoyou Gem Flower Hospital, Panjin
  - Huabei Petroleum Administration Bureau General Hospital, Renqiu
  - Tianjin People's Hospital, Tianjin
  - Tianjin Fourth Central Hospital, Tianjin
  - Wenzhou People's Hospital, Wenzhou
  - Xi'an Gaoxin Hospital, Xi'an
  - Xianyang Hospital of Yan 'an University, Xianyang
  - The Third Affiliatied Hospital of Xinxiang Medical University, Xinxiang
  - Zaozhuang Municipal Hospital, Zaozhuang
- Czechia (11):
  - Hornicka nemocnice s poliklinikou Bilina s.r.o., Bílina
  - Medicus Services SRO, Brandýs nad Labem
  - Centrum pro zdravi - kardiologie s.r.o., Brno
  - Kardiologicka ambulance Brno s.r.o., Brno
  - Cevni ambulance - MATMED s.r.o., Hodonín
  - MUDr. Tomas Edelsberger - diabetologicka ambulance, Krnov
  - KARDIOLOGIE - LIBEREC s.r.o., Liberec
  - PreventaMed s.r.o., Olomouc
  - CCR Ostrava s.r.o., Ostrava
  - CCR Czech a.s., Pardubice
  - Kardiologie COR s.r.o., Prague
- Denmark (5):
  - Aarhus University Hospital, Aarhus
  - Amager Hospital, Copenhagen S
  - Sydvestjysk Hospital, Esbjerg
  - Godstrup Regional Hospital (Gødstrup), Herning
  - Viborg Regional Hospital, Viborg
- Georgia (9):
  - Health LTD, Batumi
  - JSC Curatio, Tbilisi
  - Acad. G. Chapidze Emergency Cardiology Center LTD, Tbilisi
  - Bokhua Memorial Cardiovascular Center LTD, Tbilisi
  - Vitamedi LTD, Tbilisi
  - Medi Club Georgia LLC, Tbilisi
  - Georgian-Ducht Hospital LTD, Tbilisi
  - The First Medical Center LTD, Tbilisi
  - Adapti LTD, Tbilisi
- Japan (17):
  - Chiba University Hospital, Chiba
  - New Tokyo Heart Clinic, Chiba
  - Japan Community Health Care Organization Kyushu Hospital, Fukuoka
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Hyogo Prefectural Harima-Himeji General Medical Center, Hyōgo
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - Komatsu Municipal Hospital, Ishikawa
  - Public Central Hospital of Matto lshikawa, Ishikawa
  - Showa University Northern Yokohama Hospital, Kanagawa
  - Kokura Memorial Hospital, Kitakyushu
  - Niigata University Medical & Dental Hospital, Niigata
  - The Sakakibara Heart Institute of Okayama, Okayama
  - Sakurabashi Watanabe Hospital, Osaka
  - National Cerebral and Cardiovascular Center Research Institute, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Osaka
  - Tokyo Saiseikai Central Hospital, Tokyo
- Netherlands (20):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academic Medical Center - Department of Vascular Medicine, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Tergooiziekenhuizen Blaricum, Blaricum
  - IJsselland ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis, Delft
  - Ziekenhuis Deventer, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Martini Ziekenhuis, Groningen
  - St. Jansdal Ziekenhuis, Harderwijk
  - Canisius-Wilhelmina Ziekenhuis (CWZ), Nijmegen
  - Laurentius Hospital Roermond, Roermond
  - Bravis ziekenhuis - Locatie Roosendaal, Roosendaal
  - Ikazia Ziekenhuis, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Gelre Ziekenhuizen - Locatie Zutphen, Zutphen
  - Albert Schweitzer Ziekenhuis - Location Dordrecht, Zwijndrecht
- Poland (21):
  - Centrum Medyczne Kermed - Renata Bijata-Bronisz I Ewa Kowalinska Spólka Jawna, Bydgoszcz
  - CENTRUM MEDYCZNE INTERCOR Sp. z o.o., Bydgoszcz
  - NZOZ Twoje Zdrowie EL Sp. z o.o., Elblag
  - Indywidualna Specjalistyczna Praktyka Lekarska w Dziedzinie Kardiologii, lek. med. Krzysztof Cymerman, Gdynia
  - Silmedic Sp. z o.o., Katowice
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - FutureMeds Lodz, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Indywidualna Specjalistyczna Praktyka Lekarska Wlodzimierz Kus, Lodz
  - Clinical Best Solutions - Lublin, Lublin
  - KO - MED Centra Kliniczne Lublin II, Lublin
  - Futuremeds Olsztyn, Olsztyn
  - Ostrowieckie Centrum Medyczne spólka cywilna Anna Olech-Cudzik, Ostrowiec Świętokrzyski
  - Aka-Med Centrum Spólka Z Ograniczona Odpowiedzialnoscia, Ruda Śląska
  - Nowe Zdrowie-Ck Kieltucki i Wspolnicy Spolka Jawna, Staszów
  - Prywatny Gabinet Lekarski Jacek Gessek, Torun
  - FutureMeds Warszawa Centrum, Warsaw
  - Clinical Best Solutions Sp. z.o.o Spolka Komandytowa, Warsaw
  - FutureMeds Targowek, Warsaw
  - FutureMeds Sp. z o.o, Wroclaw
  - 4 Wojskowy Szpital Kliniczny z Poliklinika Samodzielny Publiczny ZOZ we Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicholls SJ, Nelson AJ, Ditmarsch M, Kastelein JJP, Ballantyne CM, Ray KK, Navar AM, Nissen SE, Goldberg AC, Brunham LR, Curcio D, Wuerdeman E, Neild A, Kling D, Hsieh A, Dicklin MR, Ference BA, Laufs U, Banach M, Mehran R, Catapano AL, Davidson MH. Obicetrapib on top of maximally tolerated lipid-modifying therapies in participants with or at high risk for atherosclerotic cardiovascular disease: rationale and designs of BROADWAY and BROOKLYN. Am Heart J. 2024 Aug;274:32-45. doi: 10.1016/j.ahj.2024.05.002. Epub 2024 May 4. PMID 38705341
- [Result] Nicholls SJ, Nelson AJ, Ditmarsch M, Kastelein JJP, Ballantyne CM, Ray KK, Navar AM, Nissen SE, Harada-Shiba M, Curcio DL, Neild A, Kling D, Hsieh A, Butters J, Ference BA, Laufs U, Banach M, Mehran R, Catapano AL, Huo Y, Szarek M, Balinskaite V, Davidson MH; BROADWAY Investigators. Safety and Efficacy of Obicetrapib in Patients at High Cardiovascular Risk. N Engl J Med. 2025 Jul 3;393(1):51-61. doi: 10.1056/NEJMoa2415820. Epub 2025 May 7. PMID 40337982
- [Derived] Davidson MH, Szarek M, Scheltens P, Vijverberg E, Hsieh A, Ditmarsch M, Kling D, Curcio D, Nicholls SJ, Ray KK, Cummings JL, Kastelein JJ. Effect of obicetrapib, a potent cholesteryl ester transfer protein inhibitor, on p-tau217 levels in patients with cardiovascular disease. J Prev Alzheimers Dis. 2026 Jan;13(1):100394. doi: 10.1016/j.tjpad.2025.100394. Epub 2025 Oct 17. PMID 41109840
- See also: Study design paper — https://pubmed.ncbi.nlm.nih.gov/38705341/
- See also: Study primary results paper — https://pubmed.ncbi.nlm.nih.gov/40337982/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4214 patients were screened: out of 4214, 2530 participants were randomized (2:1) (obicetrapib: placebo): 1686 participants to the obicetrapib 10 mg group and 844 participants to the placebo group
Period: Overall Study
Arm/Group | Placebo | Obicetrapib 10mg
Started | 844 | 1686
Completed | 795 | 1600
Not Completed | 49 | 86
Not completed — Lost to Follow-up | 16 | 38
Not completed — Withdrawal by Subject | 20 | 27
Not completed — Death | 11 | 17
Not completed — Physician Decision | 0 | 1
Not completed — Participant Moved Away | 0 | 2
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Population is defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Obicetrapib 10mg | Total
Number analyzed (Participants) | 844 | 1686 | 2530
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9.61) | 65.4 (9.90) | 65.4 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 573 | 853
  Male | 564 | 1113 | 1677
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 80 | 126
  Not Hispanic or Latino | 798 | 1605 | 2403
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 150 | 312 | 462
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 112 | 151
  White | 647 | 1241 | 1888
  More than one race | 2 | 7 | 9
  Unknown or Not Reported | 5 | 9 | 14
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — Measure Description: Baseline LDL-C is defined as the last measurement prior to the first dose of study drug. LDL-C was measured by Preparative Ultracentrifugation (PUC).
  mg/dL | 98.4 (37.94) | 98.1 (37.05) | 98.25 (37.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 84 [PUC]
Description: LS mean percent change from baseline to Day 84 in Low-Density Lipoprotein Cholesterol (LDL-C) in the obicetrapib group compared to the placebo group [PUC]. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 84 Days
Population: Baseline Population is defined as all participants who were randomized in the study. Baseline values were defined as last measurement prior to the first dose of study drug. Missing values were imputed using a multiple imputation model assuming the data are missing not at random. Missing measurements of non-retrieved dropouts were modeled by known measurements from retrieved dropouts in the same treatment group.
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 842 | 1679
percent change from baseline | 2.70 (1.571) | -29.94 (1.104)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -32.65, 95% CI 2-sided [-35.79 to -29.50], Standard Error of Mean 1.602

2. Secondary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol (LDL-C) From Baseline to Day 180 [Martin/Hopkins]
Description: LS mean percent change from baseline to Day 180 in Low-Density Lipoprotein Cholesterol (LDL-C) in the obicetrapib group compared to the placebo group [Martin/Hopkins]. LDL-C value was calculated using the Martin/Hopkins equation unless TG >= 400 mg/dL or LDL-C <= 50 mg/dL; where, LDL-C value was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 180 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 4.68 (1.625) | -29.09 (1.176)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -33.78, 95% CI 2-sided [-37.07 to -30.49], Standard Error of Mean 1.678

3. Secondary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol (LDL-C) From Baseline to Day 365 [PUC]
Description: LS mean percent change from baseline to Day 365 in Low-Density Lipoprotein Cholesterol (LDL-C) in the obicetrapib group compared to the placebo group [PUC]. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 365 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 842 | 1679
percent change from baseline | -1.27 (1.798) | -25.25 (1.480)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — The hierarchical testing procedure would only be conducted if the previous secondary efficacy endpoint reached a statistically significant treatment effect at p-value<0.05; Least Squares (LS) Means = -23.98, 95% CI 2-sided [-27.87 to -20.09], Standard Error of Mean 1.979

4. Secondary Outcome: Percent Change in Apolipoprotein B (ApoB) From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in apolipoprotein B (ApoB) in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 1.08 (0.911) | -17.84 (0.669)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -18.92, 95% CI 2-sided [-20.76 to -17.09], Standard Error of Mean 0.936

5. Secondary Outcome: Percent Change in Apolipoprotein B (ApoB) From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in apolipoprotein B (ApoB) in obicetrapib group compared to the placebo group.
Time Frame: 180 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 2.23 (1.033) | -16.07 (0.742)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -18.31, 95% CI 2-sided [-20.38 to -16.23], Standard Error of Mean 1.057

6. Secondary Outcome: Percent Change in Apolipoprotein B (ApoB) From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in apolipoprotein B (ApoB) in obicetrapib group compared to the placebo group.
Time Frame: 365 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | -1.77 (1.165) | -15.57 (0.914)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -13.80, 95% CI 2-sided [-16.20 to -11.41], Standard Error of Mean 1.219

7. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 2.81 (1.212) | -26.64 (0.892)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -29.44, 95% CI 2-sided [-31.89 to -26.99], Standard Error of Mean 1.251

8. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in Non-high-density Lipoprotein Cholesterol (non-HDL-C) in obicetrapib group compared to the placebo group.
Time Frame: 180 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 3.68 (1.302) | -24.63 (0.972)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -28.32, 95% CI 2-sided [-30.94 to -25.69], Standard Error of Mean 1.339

9. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in Non-high-density Lipoprotein Cholesterol (non-HDL-C) in obicetrapib group compared to the placebo group.
Time Frame: 365 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 0.63 (1.480) | -22.38 (1.186)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = -23.02, 95% CI 2-sided [-26.09 to -19.95], Standard Error of Mean 1.564

10. Secondary Outcome: Percent Change in HDL-C From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in High-density Lipoprotein Cholesterol (HDL-C) in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 0.61 (1.391) | 136.87 (1.857)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = 136.26, 95% CI 2-sided [132.46 to 140.07], Standard Error of Mean 1.939

11. Secondary Outcome: Percent Change in HDL-C From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in High-density Lipoprotein Cholesterol (HDL-C) in obicetrapib group compared to the placebo group.
Time Frame: 180 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 1.18 (1.897) | 135.61 (2.192)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = 134.43, 95% CI 2-sided [129.84 to 139.03], Standard Error of Mean 2.343

12. Secondary Outcome: Percent Change in HDL-C From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in High-density Lipoprotein Cholesterol (HDL-C) in obicetrapib group compared to the placebo group.
Time Frame: 365 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 3.36 (1.651) | 125.40 (2.193)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Least Squares (LS) Means = 122.04, 95% CI 2-sided [117.53 to 126.55], Standard Error of Mean 2.299

13. Secondary Outcome: Percent Change in Lp(a) From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Lipoprotein (a) [Lp(a)] in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 13.65 (8.240) | -0.48 (19.855)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 10mg; Test type: Superiority; p = 0.4841, ANCOVA — The hierarchical testing procedure would only be conducted if the previous secondary efficacy endpoint reached a statistically significant treatment effect at p-value<0.05; therefore hierarchical testing was stopped for subsequent secondary endpoints; Least Squares (LS) Means = -14.12, 95% CI 2-sided [-53.68 to 25.44], Standard Error of Mean 20.183

14. Secondary Outcome: Percent Change in Apolipoprotein A1 (ApoA1) From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Apolipoprotein A1 (ApoA1) in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 0.26 (0.597) | 43.44 (0.686)

15. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Total Cholesterol (TC) in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | -0.02 (0.757) | 17.66 (0.702)

16. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in Total Cholesterol in obicetrapib group compared to the placebo group.
Time Frame: 180 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 0.85 (0.893) | 18.68 (0.769)

17. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in Total Cholesterol in obicetrapib group compared to the placebo group.
Time Frame: 365 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | -0.58 (1.030) | 17.96 (0.886)

18. Secondary Outcome: Percent Change in Triglycerides From Baseline to Day 84
Description: LS mean percent change from baseline to Day 84 in Triglycerides in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 7.66 (1.814) | -0.17 (1.445)

19. Secondary Outcome: Percent Change in Triglycerides From Baseline to Day 180
Description: LS mean percent change from baseline to Day 180 in Triglycerides in obicetrapib group compared to the placebo group.
Time Frame: 180 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 8.22 (2.061) | 0.25 (1.584)

20. Secondary Outcome: Percent Change in Triglycerides From Baseline to Day 365
Description: LS mean percent change from baseline to Day 365 in Triglycerides in obicetrapib group compared to the placebo group.
Time Frame: 365 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | 6.33 (2.135) | 0.60 (1.781)

21. Post Hoc Outcome: Percent Change in Lp(a) From Baseline to Day 84 (Hodges-Lehman)
Description: Median percent change from baseline to Day 84 in Lipoprotein (a) [Lp(a)] in obicetrapib group compared to the placebo group.
Time Frame: 84 Days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 10mg
Number analyzed (Participants) | 843 | 1685
percent change from baseline | -0.9 [-15.7 to 13.0] | -32.3 [-62.8 to -4.7]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 54
Description: Safety Population included all participants who received at least 1 dose of any study drug.
Arm/Group | Placebo | Obicetrapib 10mg
All-Cause Mortality (participants affected / at risk) | 12/843 | 19/1685
Serious Adverse Events (participants affected / at risk) | 117/843 | 211/1685
Other Adverse Events (participants affected / at risk) | 241/843 | 459/1685
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=843) | Obicetrapib 10mg (N=1685)
Acute myocardial infarction (Cardiac disorders) | 10 (10) | 17 (18)
Angina unstable (Cardiac disorders) | 8 (9) | 17 (17)
Coronary artery disease (Cardiac disorders) | 4 (5) | 7 (8)
Myocardial infarction (Cardiac disorders) | 7 (8) | 3 (3)
Cardiac failure (Cardiac disorders) | 4 (4) | 5 (5)
Angina pectoris (Cardiac disorders) | 0 (0) | 7 (7)
Acute left ventricular failure (Cardiac disorders) | 4 (4) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 6 (6)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (5)
Bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (4) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 3 (3)
Chronic coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (2)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 9 (9)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4)
Cellulitis (Infections and infestations) | 0 (0) | 4 (5)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 7 (7)
Transient ischaemic attack (Nervous system disorders) | 3 (4) | 6 (7)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 7 (7)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 4 (4)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Embolic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2)
Sudden cardiac death (General disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 2 (2) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 2 (2)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Fat necrosis (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniofacial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (3) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 5 (5)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Primary hyperaldosteronism (Endocrine disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=843) | Obicetrapib 10mg (N=1685)
COVID-19 (Infections and infestations) | 48 (49) | 81 (81)
Upper respiratory tract infection (Infections and infestations) | 33 (35) | 49 (54)
Nasopharyngitis (Infections and infestations) | 22 (26) | 43 (55)
Urinary tract infection (Infections and infestations) | 21 (25) | 39 (41)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (28) | 38 (40)
Hyperglycaemia (Metabolism and nutrition disorders) | 28 (33) | 44 (46)
Headache (Nervous system disorders) | 17 (18) | 43 (45)
Dizziness (Nervous system disorders) | 15 (15) | 40 (44)
Hypertension (Vascular disorders) | 33 (33) | 82 (89)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study, whichever occurs first, Institution may publish the results of its study data. Institution and PI shall provide sponsor with an advance copy of any proposed communications at least 60 days prior and Sponsor shall have 60 days to review. Sponsor may request (a) the deletion of any Confidential Information, (b) reasonable changes, or (c) a delay for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT05142722/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT05142722/SAP_001.pdf